CLINICAL TRIAL: NCT03554538
Title: Development and Evaluation of Efficacy of a Web App With Multimedia Animations to Teach Therapeutic Exercise in Shoulder Pain Patients
Brief Title: Efficacy of a Web App With Multimedia Animations to Teach Therapeutic Exercise in Shoulder Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad Complutense de Madrid (Other)
Collaborators: Hospital Universitario Fundación Alcorcón (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CI 18/16
Record Dates: First submitted 2018-05-30; First posted 2018-06-13 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Shoulder impingement syndrome; Exercise web app; Efficacy
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: There will be two randomized groups in a controlled clinical trial. The two groups will receive the same treatment based on an evidence-based exercise program taught by a physiotherapist, and one group will use the app multimedia to improve the performance and adherence. The other group won't use the app but a pamphlet, to follow exercises at home.
Who Masked: Outcomes Assessor
Masking Description: The trial will be simple blinded because of the impossibility to blind patients nor physiotherapists to treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web app exercises (Experimental): An evidence based exercise program for the shoulder pain. Web application with multimedia animations with the tailored exercise program for each patient in this group.
  Interventions: Behavioral: Web app exercises program
- Exercises (Active Comparator): An evidence based exercise program for the shoulder pain.
  Interventions: Behavioral: Exercise program

INTERVENTIONS:
Behavioral: Web app exercises program — Exercise on an evidence based program for shoulder pain with web app animations to improve performance and adherence
  Arms: Web app exercises
Behavioral: Exercise program — Exercise on an evidence based program for shoulder pain
  Arms: Exercises

SUMMARY:
The aim of this trial is to develop and evaluate a web app to teach patients about how to correctly perform a tailored program of shoulder exercises.

The exercise program will be evidence based, and there will be two groups in the study, both exercising. The follow up will be of 6 months.

DETAILED DESCRIPTION:
The web app will consist of 3D multimedia animations (video and audio) which the patient will be able to access from any device with internet connection (cell phone included).

The trial will include patients with shoulder pain because of rotator cuff tendinopathy.

The investigators will carry on a pilot study with 100 patients randomly distributed into two groups, with 6 months follow up. Both groups will perform the same treatment, but the control group won´t use the exercise app. There will be four dependent variables: correct exercise performance, compliance degree, satisfaction with the treatment and expectations to improve with treatment. As secondary dependent variables will be analyzed pain (at rest, with movement and at night), functional disability (SPADI questionnaire), and patient´s assessment of app video characteristics (usability, utility and satisfaction) and co-interventions.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 with uni or bilateral shoulder region pain
* Being able to read and write in Spanish
* Pain for at least 3 months
* Pain intensity (in rest, activity and/or at night) of at least 3/10
* Two positive clinical sings at least from: Neer sign, Hawkins-Kennedy sign, empty can or pain arc
* Must have and use at least 3 times/week email of their own and a device with internet connection

Exclusion Criteria:

* Polyarticular or generalized pain
* Cognitive impairment
* Cancer
* Serious neurological disease
* Other shoulder pain causes
* History of main trauma
* Sings or symptoms of cervical pain (excluding upper trapezius) or cervical radiculopathy
* Apprehension sing, sulcus sing
* Passive movement limitation (but final degree in horizontal abduction or extension)
* Tendon rupture in ultrasound
* Glenohumeral arthritis in plain radiographs or calcium bigger than 5mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Correctness in exercise performance | 6 weeks
  25% of patients enrolled will be checked by video recording of 3 exercise performance, and the videos will be graded by two blinded assessors with a 6 points scale, 4 evaluating motor memory and 2 evaluating declaratory memory. Every exercise recording will be form 0 to 6, so the total score will range from 0 to 18.
Compliance degree | 6 months
  It will be measured by a simple monthly diary where the patient will have to register everyday if has done or not the exercises and the degree of pain every week. Total score will correspond to the percentage of days exercising over the total expected.
Treatment satisfaction: numerical visual scale | 6 months
  This outcome will be measured with a numerical visual scale of 11 points, where on the right will be "10" as completely satisfied, and on the left "0" absolutely unsatisfied.
Expectancy of improvement with treatment | 2 weeks
  This outcome will be measured using a modified question from the "Credibility/expectancy Questionnaire", that will be pointed on a numerical visual scale of 11 points having on the right "10" as complete recovery, and on the left "0" as "no improvement". The question that will be made is "how much improvement do you think you will reach in your limitations because of the shoulder pain?"

SECONDARY OUTCOMES:
Pain intensity: numerical scale | 6 months
  Measured with a numerical scale with 11 points. 0 means "without pain" and 10 "worst pain". A 2 points change will be the minimum relevant clinical change.
Functional limitation | 6 months
  Measured with the SPADI questionnaire adapted to spanish. Consists of 13 items, 5 evaluating pain and 8 disability. The total score ranges between 0 and 130, and the final score is a percentage. Higher scores mean a higher pain and disability degree. The minimal clinical change is 8 points. A 20 points change is needed for the patient to perceive an important change.
Evaluation of the app and videos | 3 months
  A 12 points questionnaire, referred to usability, perceived usefulness and satisfaction. It´s a Likert type scale to express agreement on each question over 5 points, from complete disagreement to complete agreement. The total score is over 0- 100.

CONTACTS AND LOCATIONS:
Overall Officials: Mariano T Flórez, PhD, Principal Investigator — Hospital Universitario Fundación Alcorcón

IPD SHARING:
Plan to Share IPD: Undecided